CLINICAL TRIAL: NCT01588483
Title: Prospective Study for the Follow-up of Aortic Diameter in Patients With Arteritis Temporalis / Giant Cell Arteritis.
Brief Title: Prospective Follow-up Study of the Aortic Diameter in Patients With Giant Cell Arteritis
Acronym: ATACT
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Daniel Blockmans, prof. dr. Daniël Blockmans, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: ATACT-study
Record Dates: First submitted 2012-04-23; First posted 2012-05-01 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Giant Cell Arteritis
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- giant cell arteritis: patients with biopsy and/or scintigraphy proven GCA

SUMMARY:
Giant cell arteritis (GCA) is the most frequent vasculitis in patients above 50 years of age. The disease has limited mortality, mostly due to the development of aortic aneurysms, leading to dissection and rupture. The probability to develop this complication is 17 x higher at the level of the thoracic aorta and 2,4 x at the level of the abdominal aorta in patients with GCA when compared with a control group. Therefore, follow-up of the aortic diameter in patients with GCA is part of good clinical practice. Previous retrospective research showed a link between FDG-uptake at the level of the thoracic aorta, on positron-emission-tomography (PET) at the time of diagnosis, and the increase of diameter and volume of the thoracic aorta during follow-up (on computed tomography (CT)).

The purpose of this prospective study is to follow-up on the aortic diameter, and to correlate these measures with FDG-PET uptake at diagnosis. Ideally, this would allow us to define a group of patients at high risk to develop an aortic aneurysm, already at the time of diagnosis.

DETAILED DESCRIPTION:
As standard care, all patients with a suspicion of GCA undergo a biopsy of the temporal artery and a PET scintigraphy to evaluate the presence of large vessel vasculitis. Patients with proven GCA on biopsy and/or scintigraphy undergo a computed tomography (CT) of the aorta without the administration of contrast, at diagnosis and yearly thereafter (every 12 +/- 3 months) for 10 years.

Measurements include the diameter of the ascending aorta, aortic arch, descending aorta, suprarenal, juxtarenal and infrarenal aorta, and the volume of the thoracic and the abdominal aorta. These measurements are correlated with FDG-uptake at the level of the aorta on PET-scintigraphy at the time of diagnosis. All patients will be treated according to accepted guidelines and standard care in our center (methylprednisolone started at 32 mg/day, with slowly declining doses until stop after 1 to 1,5 years of treatment).

ELIGIBILITY:
Inclusion Criteria:

* patients with a first episode of biopsy and/or scintigraphy proven giant cell arteritis
* patients with a previous diagnosis of giant cell arteritis, in whom a yearly computed tomography of the aorta is available can opt to participate in this study
* informed consent form has to be signed by all patients

Exclusion Criteria:

* patients already treated with steroids before performance of PET-scintigraphy
* earlier episodes of giant cell arteritis, without documentation of the aortic diameter at that moment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Proven Giant Cell Arteritis
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Diameter of aorta. | yearly, until 10 years after diagnosis
  diameter of ascending aorta, arcus aortae, descending aorta, suprarenal, juxtarenal and infrarenal abdominal aorta
Volume of aorta | yearly, until 10 years after diagnosis
  volume of the thoracic and abdominal aorta

CONTACTS AND LOCATIONS:
Overall Officials: Daniël Blockmans, MD, PhD, Principal Investigator — University Hospital, Gasthuisberg
Locations (1):
- University Hospital Leuven, Leuven, Belgium

REFERENCES:
- [Background] Blockmans D, Coudyzer W, Vanderschueren S, Stroobants S, Loeckx D, Heye S, De Ceuninck L, Marchal G, Bobbaers H. Relationship between fluorodeoxyglucose uptake in the large vessels and late aortic diameter in giant cell arteritis. Rheumatology (Oxford). 2008 Aug;47(8):1179-84. doi: 10.1093/rheumatology/ken119. Epub 2008 May 31. PMID 18515868